CLINICAL TRIAL: NCT03080532
Title: Diet Interactions With Human Gut Microbiota. The Potential Role of Mediterranean Diet Adherence. DIAGRAM, a Pilot Study
Acronym: DIAGRAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); Mediterranean Agronomic Institute of Chania (MAICh) - CIHEAM, Greece (Unknown); Neuromed IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0278; 2016-A00421-49 (Other: 2016-A00421-49)
Record Dates: First submitted 2016-09-09; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Human Gut Microbiota
Keywords: Microbiome; Mediterranean diet

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- european population
  Interventions: Other: dietary habits

INTERVENTIONS:
Other: dietary habits

SUMMARY:
Despite the strong evidence on health benefits of traditional MeD, not many studies have broadly and systematically been made for the potential role and relationship of the MeD in the composition of the gut microbiota.

Furthermore, little is known about the composition of the gut microbiota in individuals with defined dietary habits on the Mediterranean pattern.

This work is aiming at comparatively studying the gut microbiota of three different dietary oriented european populations. In particular, biological samples and related information will be collected from populations with high adherence to Mediterranean diet (MeD) in Crete - Greece and Molise region - Italy. These data will be comparatively assessed with those provided by a sample population with high adherence to Western diet in Auvergne - France.

DETAILED DESCRIPTION:
All the participants will give freely their written informed consent before their selection in the study.

Information on demographics, anthropometrics, vital signs, relevant medical history and concomitant medication, dietary habits, usual dietary intake and nutritional supplements will be collected. Habitual physical activity will be performed using the short form of the IPAQ survey. All inclusion and exclusion criteria will be checked by the investigator or co-investigator.

All selected volunteers will be asked to maintain their usual dietary habits and continue their normal physical habits. All volunteers will complete a follow-up questionnaire to obtain information about any changes in medication use, disease etc.

All selected volunteers will collect one stool sample and will complete two 24h dietary recalls, and questionnaires related to digestive function and life style.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 to 60 years
* Healthy (apparently free of diseases)
* Moderately physically active
* Habitually eating foods representative of their community (Cretan diet, Italian Mediterranean diet, French Auvergnat diet). The assessment of the consumption of such food will be based to a detailed dietary history retrieved by a nutrition specialist)

Exclusion Criteria:

* Following any kind of treatment, notably antibiotics the last 3 months
* Sedentary lifestyle
* BMI <18.5 Kg/m2-or >27Kg/m2
* Smokers
* Excessive alcohol consumption (>3 glasses/d for men and >2 glasses/d for women)
* To be frequent travelers, particularly to overseas destinations
* Pregnant or women at lactation
* Individual unable to give informed consent or refusing to sign informed consent

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: european populations
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-02 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Bacterial species composition of the fecal microbiota | at day 1

SECONDARY OUTCOMES:
Beta diversity of fecal microbiota | at day 1
Core microbiota (Alpha and Beta diversity of samples) | at day 1
  Taxonomic affiliation will be performed after clustering of sequences at 97% to bacterial/archaeal groups using referenced databases: GreenGenes-RDP. Alpha and Beta diversity of samples will be determined after normalization of sample size. Analyses will also determine the core microbiota of each Group.

CONTACTS AND LOCATIONS:
Overall Officials: Ruddy RICHARD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France